CLINICAL TRIAL: NCT02964195
Title: Efficacy of Rifaximin in Treatment of Cirrhotic Gastroesophageal Variceal Hemorrhage: A Multi-center Randomized Controlled Clinical Trial
Brief Title: Efficacy of Rifaximin in Treatment of Cirrhotic Gastroesophageal Variceal Bleeding
Acronym: EoR-GEVB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Lanzhou University Second Hospital (Other); Beijing Ditan Hospital (Other); Shandong Provincial Hospital (Other Government); Renmin Hospital of Wuhan University (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Principal Investigator, Shiyao Chen, Professor, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CSY-Rifaximin-HXQ
Record Dates: First submitted 2016-11-07; First posted 2016-11-16 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Cirrhosis; Esophageal and Gastric Varices; Gastrointestinal Hemorrhage
MeSH Terms: conditions — Fibrosis; Esophageal and Gastric Varices; Gastrointestinal Hemorrhage | interventions — Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rifaximin Group (Experimental): Rifaximin 400 mg bid for 2 month,
  Interventions: Drug: Rifaximin
- Control (No Intervention): Routine endoscopic treatment without prophylactic use of antibiotics

INTERVENTIONS:
Drug: Rifaximin — ALFA WASSERMANN S.p.A.
  Other Names: XIFAXAN
  Arms: Rifaximin Group

SUMMARY:
The purpose of the study is to evaluate the efficacy of Rifaximin in the treatment of cirrhotic gastroesophageal variceal bleeding.

DETAILED DESCRIPTION:
Gastroesophageal variceal bleeding is the most common and life-threatening condition in patients with portal hypertension, which are susceptibility to bacterial infection. However, the prophylaxis use of antibiotics remained uncertain and lack of high level evidences.

The purpose of the study is to evaluate the efficacy of Rifaximin in the treatment of cirrhotic gastroesophageal variceal bleeding.

ELIGIBILITY:
Inclusion Criteria:

* 18 y.o. ≤age≤75 y.o.;
* Cirrhotic gastroesophageal variceal bleeding underwent endoscopic treatment (include esophageal varices ligation, endoscopic injection sclerosis and gastric N-butyl-cyanoacrylate injection).

Exclusion Criteria:

* age <18 y.o. or age > 75 y.o.;
* Never had the variceal bleeding episode before;
* Do not have endoscopic treatment;
* combined with other malignant tumor (not exclude patients with hepatocellular carcinoma who don't not need treatment at the moment);
* Known infection after endoscopic treatment (Fever, microbial cultures positive, et al.)
* Massive ascites or combined with other high risk factor that require prophylaxis use of antibiotics.
* Acute variceal bleeding within 5 days.
* Use of other antibiotics in the past 2 weeks;
* Refuse to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-10 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
All clinical events | 8 weeks
  All clinical events were defined as occurrence rebreeding, ascitic fluid infection, hepatorenal syndrome, hepatopulmonary syndrome, portal vein thrombosis, or death.

SECONDARY OUTCOMES:
All clinical events | 6 months
  All clinical events were defined as occurrence rebreeding, ascitic fluid infection, or death.
Serum endotoxin, | 8 weeks, and 6 months
coagulation function | 8 weeks, and 6 months
inflammatory factors including IL-6, IL-8, TNF-a, IL-1beta | 8 weeks, and 6 months
Glucose breath hydrogen test | 8 weeks, and 6 months
changes of intestinal flora | 8 weeks, and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Shiyao CHEN, M.D., Principal Investigator — Zhongshan Hospital, Fudan University, Shanghai
Locations (1):
- 180 Fenglin Road, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bass NM, Mullen KD, Sanyal A, Poordad F, Neff G, Leevy CB, Sigal S, Sheikh MY, Beavers K, Frederick T, Teperman L, Hillebrand D, Huang S, Merchant K, Shaw A, Bortey E, Forbes WP. Rifaximin treatment in hepatic encephalopathy. N Engl J Med. 2010 Mar 25;362(12):1071-81. doi: 10.1056/NEJMoa0907893. PMID 20335583
- [Background] Garcia-Tsao G, Sanyal AJ, Grace ND, Carey W; Practice Guidelines Committee of the American Association for the Study of Liver Diseases; Practice Parameters Committee of the American College of Gastroenterology. Prevention and management of gastroesophageal varices and variceal hemorrhage in cirrhosis. Hepatology. 2007 Sep;46(3):922-38. doi: 10.1002/hep.21907. No abstract available. PMID 17879356
- [Background] Gasbarrini A, Corazza GR, Gasbarrini G, Montalto M, Di Stefano M, Basilisco G, Parodi A, Usai-Satta P, Vernia P, Anania C, Astegiano M, Barbara G, Benini L, Bonazzi P, Capurso G, Certo M, Colecchia A, Cuoco L, Di Sario A, Festi D, Lauritano C, Miceli E, Nardone G, Perri F, Portincasa P, Risicato R, Sorge M, Tursi A; 1st Rome H2-Breath Testing Consensus Conference Working Group. Methodology and indications of H2-breath testing in gastrointestinal diseases: the Rome Consensus Conference. Aliment Pharmacol Ther. 2009 Mar 30;29 Suppl 1:1-49. doi: 10.1111/j.1365-2036.2009.03951.x. PMID 19344474
- [Background] Hwang JH, Shergill AK, Acosta RD, Chandrasekhara V, Chathadi KV, Decker GA, Early DS, Evans JA, Fanelli RD, Fisher DA, Foley KQ, Fonkalsrud L, Jue T, Khashab MA, Lightdale JR, Muthusamy VR, Pasha SF, Saltzman JR, Sharaf R, Cash BD; American Society for Gastrointestinal Endoscopy. The role of endoscopy in the management of variceal hemorrhage. Gastrointest Endosc. 2014 Aug;80(2):221-7. doi: 10.1016/j.gie.2013.07.023. No abstract available. PMID 25034836
- [Background] Vlachogiannakos J, Viazis N, Vasianopoulou P, Vafiadis I, Karamanolis DG, Ladas SD. Long-term administration of rifaximin improves the prognosis of patients with decompensated alcoholic cirrhosis. J Gastroenterol Hepatol. 2013 Mar;28(3):450-5. doi: 10.1111/jgh.12070. PMID 23216382